CLINICAL TRIAL: NCT00327613
Title: Plasma Levels of Matrix Metalloproteinases and Degree of DNA Fragmentation in Patients With Pseudoexfoliation Syndrome and Open-Angle Glaucoma (PEXG)
Brief Title: Plasma Levels of Matrix Metalloproteinases (MMPs) and Degree of DNA Fragmentation in Pseudoexfoliation (PEX) Glaucoma
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Selim Orgul, University Hospital, Basel, Switzerland
Other Study IDs: 066-WUK-2005-001
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Pseudoexfoliation Syndrome; Glaucoma
Keywords: PEX; glaucoma; MMP; DNA degradation; POAG; Healthy subjects
MeSH Terms: conditions — Exfoliation Syndrome; Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Glaucoma is a worldwide leading cause of blindness. The key feature of this ocular neuropathy is characterized by an excavating optic nerve head. Loss of retinal ganglion cells is the final end point in blinding diseases of the optic nerve such as glaucoma. It is known that neuronal cell death in glaucoma occurs by apoptotic mechanism. In earlier studies, the investigators demonstrated that the process of apoptosis is reflected in circulating leukocytes by different parameters, like differential messenger ribonucleic acid (mRNA) expression and an increased fragmentation of the deoxyribonucleic acid (DNA). Such alterations point out a relationship between cellular stress and apoptotic events.

Based on the results of mRNA-expression, the investigators also expect alterations on the protein level.

This study is, therefore, designed to characterize the proteome related to the proteins involved in cell death related pathways.

Thus the expression pattern of several proteins in leukocytes from patients with primary open angle glaucoma will be analyzed by techniques like Western-blot and tandem mass spectrometry. These samples will be compared with healthy controls. In addition, they will be also compared with samples from patients with Parkinson's disease. Since glaucoma is a neurodegenerative disease, these patients will be included as a positive control in this study.

DETAILED DESCRIPTION:
Hypothesis:

Subjects with pseudoexfoliation syndrome in combination with glaucoma may have an altered activity of plasma matrix-metalloproteinase activity and a higher degree of DNA fragmentation in the leukocytes.

Specific aims:

Determination of the level of plasma matrix-metalloproteinase activity and of the degree of DNA fragmentation of leukocytes in patients with pseudoexfoliation syndrome glaucoma (PEX) in comparison to patients with primary open angle glaucoma (POAG).

Background:

One of the main pathogenic factors for the development of glaucoma is an increased intraocular pressure (IOP), which leads to a direct or indirect damage of the nerve fibers in the area of the optic disk. The raise of IOP is based on the increased outflow resistance of the trabecular meshwork due to an excessive accumulation of extracellular material in the juxtacanalicular tissue of the meshwork in eyes with primary open-angle glaucoma (POAG), and an impaired turnover of the trabecular meshwork matrix, which is of paramount importance to the regulation and maintenance of aqueous humor outflow.

Pseudoexfoliation (PEX) syndrome is a systemic disorder of the extracellular matrix, which represents the most common identifiable cause of open-angle glaucoma. There is increasing evidence suggesting that PEX syndrome may be a type of fibrosis associated with excessive synthesis and deposition of an abnormal elastic fibrillar material in many intra- and extraocular tissues. Active involvement of the trabecular meshwork in this abnormal matrix process leading to progressive accumulation of PEX material in the juxtacanalicular tissue is considered to be the primary cause of chronic pressure elevation in eyes with PEX syndrome. However, the mechanisms responsible for this aberrant matrix process remain unknown. Excessive production and accumulation of abnormal matrix components may be due to increased de-novo synthesis, decreased turnover of matrix components, or both.

Extracellular matrix turnover is mediated by matrix metalloproteinases (MMPs), a large family of endopeptidases with variable substrate spectra, the presence of which has been described in human aqueous humor.

The activity of these enzymes is regulated in part by specific endogenous inhibitors, the tissue inhibitors of metalloproteinases (TIMPs). Dysregulated expression of MMPs and TIMPs has been implicated in many disease processes accompanied by abnormal matrix production, such as fibrotic disorders, and a variety of other disease states. In the eye, abnormal expression of MMPs has been implicated, among many other disorders, in glaucoma, in proliferative vitreoretinopathy, secondary cataract formation, and the pathogenesis of pterygia. Therefore, MMPs and TIMPs are likely candidates to be involved in the abnormal extracellular matrix metabolism characteristic of PEX syndrome/glaucoma (PEXG) and POAG.

PEX seems to be an independent risk factor for glaucoma. Possibly, this may be due to an altered perfusion. So, PEX syndrome represents not only the most common identifiable cause of open-angle glaucoma, but also a risk factor for cardiovascular diseases. PEX syndrome and iris trans-illumination defects are seen in patients with transient ischemic attacks. At the microcirculatory level, ischemia/reperfusion (I/R) injury is thought to be initiated by chemotactic accumulation of circulating leukocytes, their activation and interaction with the endothelium of postcapillary venules. In addition, oxygen free radicals are thought to play a pivotal role in the pathogenesis of I/R injury. A variety of experimental models of ischemic injury have shown that free radicals induce post-ischemic oxidative damage to DNA. Although several human studies have revealed that oxygen radicals generated by other mechanisms like irradiation, only few data exist that demonstrate the influence of reperfusion-associated oxygen radicals on DNA in humans. We hypothesize that the pathogenic processes in PEX may be reflected in leukocytes.

Depending on the results that glaucoma patients differ on the level of their mRNA expression for various MMPs in peripheral leukocytes and that PEX syndrome is often seen with transient ischemic attacks, we assume differences in the activity of MMPs in the plasma as well as changes in the DNA stability in peripheral leukocytes of patients with PEX glaucoma.

This study is, therefore, designed to analyze the activity of gelatinases (MMP-2 and -9) in plasma and the degree of DNA fragmentation in peripheral leukocytes of patients with PEX syndrome and PEXG compared to POAG and controls.

ELIGIBILITY:
Inclusion Criteria:

* German native speakers
* Age between 18-80 years
* Pseudoexfoliation syndrome
* Pseudoexfoliation syndrome with open-angle glaucoma
* Primary open-angle glaucoma

Exclusion Criteria:

* Any history of ocular or systemic diseases other than glaucoma or of drug or alcohol abuse.
* Any condition potentially interfering with the visual field results. Visual fields will be obtained from the chart.
* Any mentally impaired patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pseudoexfoliation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2005-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orgül, MD, Study Director — University Hospital, Basel, Switzerland
Locations (1):
- University Eye Clinic Basel, Basel, Canton of Basel-City, Switzerland